CLINICAL TRIAL: NCT04678882
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel-group Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Dupilumab Compared to Placebo in Japanese Patients With Atopic Dermatitis Aged 6 Months to <18 Years Whose Disease is Not Adequately Controlled With Existing Therapies
Brief Title: Dupilumab in Japanese Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC16823; U1111-1301-1257 (Registry Identifier: ICTRP); 2020-002601-26 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Double dose on day1 and followed by single dose every 2 weeks or single dose every 4 weeks
  Interventions: Drug: Dupilumab SAR231893
- Placebo (Placebo Comparator): Double dose on day1 and followed by single dose every 2 weeks or single dose every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous (SC)
  Arms: Placebo
Drug: Dupilumab SAR231893 — Pharmaceutical form: solution for injection Route of administration: subcutaneous (SC)
  Arms: Dupilumab

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab administered concomitantly with topical corticosteroids (TCS)

Secondary Objective:

To evaluate the efficacy of dupilumab administered concomitantly with TCS. To assess the safety of dupilumab over 16 weeks of treatment when administered concomitantly with TCS in participants.

To assess immunogenicity as determined by the incidence, titer, and clinical impact of treatment-emergent anti-drug antibodies (ADA) to dupilumab over time in pediatric patients with atopic dermatitis (AD) (aged ≥6 months to <18 years old) To assess the concentration of dupilumab in serum following administration concomitantly with TCS.

DETAILED DESCRIPTION:
For participant who declines to enter open-lebal extension (OLE), the duration of the study for each participant is approximately 33 weeks (including screening and follow-up) For participant choosing enter OLE, the duration is approximately 21 weeks (including screening) plus 3 years OLE period or until approval of the indication in Japan whichever is sooner.

ELIGIBILITY:
Inclusion criteria :

Japanese and ≥6 months to <18 years of age, at the time of signing the informed consent and/or assent.

Diagnosis of AD according to the American Academy of Dermatology consensus criteria at screening visit.

Chronic AD diagnosed at least 1 year prior to the screening visit (for participants between 6 months to <1 year of age, the requirement is to have had chronic AD for 3 months).

(Investigator's Global Assessment) IGA ≥ 3 at screening and baseline visits. (Eczema Area and Severity Index) EASI ≥16 at screening and baseline visits. Baseline peak pruritus Numerical Rating Scale (NRS) average score for maximum itch intensity ≥4 for participants ≥12 to <18 years of age.

Baseline worst itch NRS or worst scratch/itch NRS weekly average score for maximum itch or scratch/itch intensity ≥4 for participants ≥6 months to <12 years of age.

Body surface area (BSA) of AD involvement >10% at screening and baseline visits.

With documented recent history (within 6 months before the baseline visit) of inadequate response to topical AD medication(s).

At least 11 (of a total of 14) applications of a stable dose of topical emollient (moisturizer) twice daily immediately before the baseline visit.

Willing and able to comply with all clinic visits and study-related procedures. Participant, either alone or with help of parents/legal guardians (for 6 years old to less than18 years of age) or parents/caregiver or legal guardians (for 6 months to less than 6 years of age) as appropriate, must be able to understand and complete study-related questionnaires.

Body weight ≥5 kg at baseline. Contraceptive use by female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion criteria:

Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the baseline visit or during the screening period.

Known or suspected immunodeficiency, including history of invasive opportunistic infections Participants with active tuberculosis (TB) or non-tuberculous mycobacterial infection, or a history of incompletely treated TB will be excluded from the study unless it is well documented by a specialist that the participant has been adequately treated and can now start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist.

Known history of human immunodeficiency virus (HIV)-1 and HIV-2 infection or HIV seropositivity at the screening

Participants with any of the following result at the screening:

* Positive (or indeterminate) Hepatitis B surface antigen (HBs Ag) or,
* Positive hepatitis B core antibody (HBc Ab) confirmed by positive hepatitis B virus (HBV) DNA or,
* Positive hepatitis C antibody (HCV Ab) confirmed by positive hepatitis C virus (HCV) RNA.

Presence of skin comorbidities that may interfere with study assessments History of malignancy within 5 years before the baseline visit History of systemic hypersensitivity or anaphylaxis to dupilumab or any other biologic therapy.

Known or suspected alcohol and/or drug abuse. Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection.

Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study.

Participant with any other medical or psychological condition including relevant laboratory or electrocardiogram (ECG) abnormalities at screening Exposure to another systemic or topical investigative drug within a certain time period prior to Visit 1 (screening), Having used any of immunosuppressive/immunomodulating drugs and phototherapy within 4 weeks before the screening visit.

Past Treatment with biologics as follows:

* Any cell-depleting agents within 6 months before the screening visit.
* Anti-IgE therapy within 4 months before the screening visit.
* Other monoclonal antibodies (which are biological response modifiers): within 5 half-lives (if known) or 16 weeks before the screening visit (Visit 1), whichever is longer.

History of important side effects to medium potency TCS Treatment with a live (attenuated) vaccine within 4 weeks before the baseline visit.

Either intravenous immunoglobulin therapy and/or plasmapheresis within 30 days prior to screening visit.

Planned or anticipated use of any prohibited medications and procedures during screening and study treatment period.

Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period Participation in a prior dupilumab clinical study or have been treated with commercially available dupilumab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Eczema Area and Severity Index (EASI)-75 (≥75% improvement from baseline EASI) | At Week 16
  The EASI is a composite index with scores ranging from 0 to 72.Higher scores indicates worse condition

SECONDARY OUTCOMES:
Percent change in EASI score | From baseline to week 16
  The EASI is a composite index with scores ranging from 0 to 72.Higher scores indicates worse condition
Percent change in weekly average of daily worst itch numerical rating scale (NRS) for participants aged ≥6 years to <12 years old | From baseline to week 16
  The worst itch NRS is a simple assessment tool those participants ≥6 years old to <12 years old will use to report the intensity of their pruritus (itch). This is an 11-point scale (0 to 10) in which 0 indicates no itching while 10 indicate worst itching possible.
Proportion of participants with Investigator's Global Assessment (IGA) 0 or 1 | At Week 16
  The IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe)
Percent change in weekly average of daily worst peak pruritus NRS for participants aged ≥12 years to <18 years old | From baseline to week 16
  The peak pruritus NRS is a simple assessment tool that participants ≥ 12 to <18 years old will use to report the intensity of their pruritus (itch) ranges from 0 to 10 with 0 being 'no itch' and 10 being the' worst itch imaginable'
Percent change in weekly average of daily worst scratch/itch NRS for participants aged ≥6 months to <6 years old | From baseline to week 16
  The worst scratch/itch NRS is a simple assessment tool those participants ≥6 years old to <6 years old range from 1 to 10 in which 0 indicates no itching while 10 indicate worst itching possible
Percent change for intensity of pruritus | From baseline to week 16
  The intensity is assessed by numerical rating scale ranging from 0 to 10 which higher scale indicate worse itch condition
Proportion of participants with EASI-50 (≥50% improvement from baseline) | At Week 16
  The EASI is a composite index with scores ranging from 0 to 72.Higher scores is worse condition
Proportion of participants with EASI-90 (≥90% improvement from baseline) | At Week 16
  The EASI is a composite index with scores ranging from 0 to 72.Higher scores is worse condition
Change in percent body surface area (BSA) affected by atopic dermatitis (AD) | From baseline to week 16
  BSA affected by atopic dermatitis will be assessed for each major section of the body (head, trunk, arms, and legs).
Change in Children's Dermatology Life Quality Index (CDLQI) (≥4 years) | From baseline to week 16
  The CDLQI is a validated questionnaire designed to measure the impact of skin disease on the Quality of Life. The higher the score, the greater the impact is on the quality of life
Change in Infants' Dermatitis Quality of Life Index (IDQOL) (<4 years) | From baseline to week 16
  The IDQOL is a validated questionnaire developed to measure the impact of skin disease on the QOL of infants and preschool children <4 years of age wil completed by the child's parent or caregiver. The higher the score, the greater the impact is on the quality of life. -
Change in Patient Oriented Eczema Measure (POEM) | From baseline to week 16
  The POEM is a 7-item (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) questionnaire used to assess disease symptoms with a scoring system of 1 to 28. The higher score, the higher morbidity
Change in weekly average of daily worst peak pruritus NRS for participants aged ≥12 years to <18 years old | From baseline to week 16
  The peak pruritus NRS is a simple assessment tool that participants ≥ 12 to <18 years old will use to report the intensity of their pruritus (itch) ranges from 0 to 10 with 1 being 'no itch' and 10 being the' worst itch imaginable'
Change in weekly average of daily worst itch NRS for participants aged ≥6 years to <12 years old | From baseline to week 16
  The worst itch NRS is a simple assessment tool those participants ≥6 years old to <12 years old range from 1 to 10 in which 1 indicates no itching while 10 indicate worst itching possible -
Change in weekly average of daily worst scratch/itch NRS for participants aged ≥6 months to <6 years old | From baseline to week 16
  The worst scratch/itch NRS is a simple assessment tool those participants ≥6 years old to <12 years old range from 1 to 10 in which 1 indicates no itching while 10 indicate worst itching possible
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), Serious Adverse Events (SAEs), and Adverse Event of Special Interest (AESI) From Baseline to 16 Weeks of Treatment | Baseline (Day 1) to Week 16
Number of Participants With Skin-Infection TEAEs (Excluding Herpetic Infections) From Baseline to 16 Weeks of Treatment | Baseline (Day 1) to Week 16
Number of Participants With TEAEs, SAEs, and AESI From Baseline of open-label extension (OLE) Through the Last Study Visit | Week 16 to Week 116
Number of Participants With Treatment-emergent Anti-drug Antibody (ADA) to Dupilumab Over Time in Pediatric Participants with AD (Aged ≥6 Months to <18 Years old) | Baseline (Day 1) to Week 116
Serum Concentration of Dupilumab up to Week 116 | Pre-dose at Baseline (Day 1), and Weeks 4, 12, 16, 24, 32, 52, 68, 92, and 116

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- Japan (19):
  - Investigational Site Number : 3920011, Nagoya, Aichi-ken
  - Investigational Site Number : 3920014, Toyoake-shi, Aichi-ken
  - Investigational Site Number : 3920015, Fukutsu-shi, Fukuoka
  - Investigational Site Number : 3920001, Hiroshima, Hiroshima
  - Investigational Site Number : 3920013, Sapporo, Hokkaido
  - Investigational Site Number : 3920009, Sapporo, Hokkaido
  - Investigational Site Number : 3920008, Kobe, Hyōgo
  - Investigational Site Number : 3920007, Kobe, Hyōgo
  - Investigational Site Number : 3920003, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 3920017, Yokohama, Kanagawa
  - Investigational Site Number : 3920010, Yokohama, Kanagawa
  - Investigational Site Number : 3920006, Tsu, Mie-ken
  - Investigational Site Number : 3920020, Sakai-shi, Osaka
  - Investigational Site Number : 3920019, Toyonaka-shi, Osaka
  - Investigational Site Number : 3920016, Kumagaya-shi, Saitama
  - Investigational Site Number : 3920023, Chuo-ku, Tokyo
  - Investigational Site Number : 3920012, Koto-ku, Tokyo
  - Investigational Site Number : 3920022, Toshima-ku, Tokyo
  - Investigational Site Number : 3920021, Habikino-shi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: 2020-002601-26 EudraCT results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2020-002601-26/results
- See also: EFC16823 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25256&tenant=MT_SNY_9011